CLINICAL TRIAL: NCT02484417
Title: A Phase I Study of Respiratory Syncytial Virus Human Challenge in Healthy Adult Volunteers
Brief Title: Respiratory Syncytial Virus Human Challenge in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 150148; 15-I-0148
Record Dates: First submitted 2015-06-25; First posted 2015-06-29 (Estimated); Last update posted 2025-04-08 (Actual); Status verified 2025-04-04

CONDITIONS: Upper Respiratory Tract Infection
Keywords: Neutralizing Antibody; Viral Shedding; Challenge; RSV; Healthy Volunteer
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1: RSV A2 10^5 PFU/dose (Experimental): Challenge 4 subjects with low dose and proceed to larger cohort after safety review.
  Interventions: Biological: RSV A2
- Cohort 2: RSV A2 10^5 PFU/dose (Experimental): Challenge 12 subjects with the low dose and proceed to high dose after safety review.
  Interventions: Biological: RSV A2
- Cohort 3: RSV A2 10^6.3 PFU/dose (Experimental): Challenge 12 subjects with the high dose
  Interventions: Biological: RSV A2

INTERVENTIONS:
Biological: RSV A2 — Intranasal inoculation of healthy volunteers with 10^5 or 10^6.3 plaque forming units (PFU) of RSV A2.

SUMMARY:
Background:

- Respiratory syncytial virus (RSV) can cause respiratory infections. Some of these can be life-threatening, especially in young children, the elderly, and people with weak immune systems. Researchers want to study RSV infection in a hospital setting in healthy adults. They want to use what they learn to test new treatments or vaccines in the future.

Objectives:

- To study how the body responds to RSV.

Eligibility:

- Healthy volunteers ages 18-50

Design:

* Participants will be screened under another protocol.
* Participants will have:
* Medical history
* Physical exams
* EKG. Heart rhythm is measured with small sticky patches on the chest, arms, and legs.
* Chest x-ray
* Pulmonary function tests. This measures how much air a person can move into and out of the lungs.
* Blood and urine tests
* Nasal washes and/or nasal swabs. For the wash, the nose will be rinsed with a sterile liquid. For the swab, the inside of the nostril will be rubbed with a cotton swab.
* Participants will have two, possibly three, follow-up outpatient visits, approximately 1, 2 and 6 months after receiving the dose of RSV.
* Participants will stay in the hospital under isolation for 7 or more days after getting the virus.
* The average stay is 10 days. Participants cannot leave the isolation unit. They cannot have visitors.
* The virus should cause a mild to medium cold.
* Participants will fill out a symptom card every day in the hospital and for 1 month after.
* Participants will have 2 follow-up visits, 28 and 56 days after leaving the hospital.
* Female participants who are sexually active must remain abstinent or use an effective form of birth control for 1 month before and after getting the virus.

DETAILED DESCRIPTION:
Respiratory syncytial virus (RSV) is the leading cause of pediatric lower respiratory tract infection. RSV also causes lower respiratory tract disease in the elderly and life-threatening disease in immunocompromised hosts. An RSV monoclonal antibody (palivizumab) is currently available for passive immunoprophylaxis in high-risk infants. Vaccines and antiviral agents are under development for the treatment and prevention of RSV, but none are licensed. The ability to challenge healthy volunteers with RSV could rapidly facilitate efficacy studies of future antivirals and vaccines. In addition, challenge studies would provide critical information on viral pathogenesis, including types of cells infected, mucosal and systemic immune response, and alterations in respiratory microbiota. Clinical trial material for human challenge studies has been prepared from live recombinant (complementary DNA-derived) RSV of subgroup A (RSV A2).

This study will be a phase 1 study in healthy adult male and non-pregnant female subjects 18 years to 50 years of age. The purpose of the trial is to define safety profiles and estimate illness rates for subjects given 2 different doses of RSV A2 challenge virus. If RSV A2 is found to be sufficiently infectious in adults, then it may be used as a challenge virus in future studies evaluating the protective efficacy of RSV vaccines or antivirals and in studies of pathogenesis of RSV.

Subjects will be admitted to the NIH Clinical Center and receive a single intranasal dose of RSV A2 at either 10^5 or 10^6.3 PFU. Subjects will remain at the Clinical Center for approximately 9-12 days for clinical evaluation. Research procedures conducted on blood and nasal swab and wash samples will include lymphocyte phenotyping, cytokine analysis, transcriptosome profiling, RSV-specific immunoglobin analysis (circulating IgG and nasal secretory IgA), quantitative viral titers and viral culture, and nasal microbiome analysis. Subjects will be discharged when their NP wash RSV results are negative for two consecutive days and they do not have any signs or symptoms suggestive of possible RSV-associated lower respiratory tract disease. Subjects will return for followup evaluation 28 and 56 days after viral challenge.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age 18-50 years.
  2. General good health, without significant medical illness, physical exam findings, or significant laboratory abnormalities as determined by the investigator.
  3. Willingness to stay confined to the inpatient unit for required study duration.
  4. Willingness to have samples stored for future research.
  5. Subjects must be of non-childbearing potential (i.e., either surgically sterilized [bilateral oophorectomy, bilateral tubal ligation, hysterectomy] or, if of child-bearing potential and sexually active with a partner who can get them pregnant, then they must be have in place an effective method of contraception for at least 30 days prior to administration of the challenge virus and until 30 days after challenge virus administration:
* intrauterine device (IUD) or equivalent
* hormonal contraceptives (e.g., consistent, continuous use of contraceptive pill, patch, ring, implant or injection)
* if participant uses contraceptive pill, patch or ring, two methods of contraception are required; a barrier method is to be used at the time of potentially reproductive sexual activity (e.g. male/female condom, cap, or diaphragm plus spermicide)
* be in a monogamous relationship with a partner who has undergone a vasectomy at least 6 months prior to first dose of study agent.

EXCLUSION CRITERIA:

The presence of any one of the following criteria is sufficient to exclude a prospective subject from enrolling in this study:

1. Female subject is pregnant or lactating OR planning to become pregnant in the timeframe that begins 30 days prior to the inoculation and ends 30 days after inoculation.
2. Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, hematologic, rheumatologic, endocrine, autoimmune, or renal disease.
3. Complete blood count (CBC), AST, ALT, or creatinine values are both outside of the NIH Department of Laboratory Medicine normal reference range and deemed clinically significant by the PI.
4. Behavioral or cognitive impairment or psychiatric disease that in the opinion of the investigator affects the ability of the subject to understand and cooperate with the study protocol.
5. A medical, occupational, or family problem as a result of alcohol or illicit drug use during the past 12 months.
6. Routine smoker of a tobacco product or marijuana currently or in the past year.
7. Current alcohol abuse or addiction.
8. Current illicit drug abuse or addiction.
9. Presence of any febrile illness or symptoms suggestive of a viral respiratory infection within 2 weeks prior to inoculation accompanied by a positive multiplex FilmArray PCR performed on nasal wash.
10. Use of corticosteroids (including nasal preparations) or immunosuppressive drugs within 30 days before inoculation.
11. A history of asthma within the past 10 years, or a current diagnosis of asthma or reactive airway disease associated with exercise, seasonal hay fever or allergic rhinitis.
12. Positive FDA-approved HIV test result prior to inoculation.
13. Positive serology for hepatitis C virus within 6 months prior to inoculation.
14. Presence of hepatitis B surface antigen within 6 months prior to inoculation.
15. A known immunodeficiency syndrome.
16. Receipt of a licensed vaccine within 4 weeks prior to viral inoculation.
17. Receipt of blood or blood-derived products (including immunoglobulin) within 6 months prior to viral inoculation. Receipt of packed red blood cells given for an emergent indication in an otherwise healthy person, and not required as ongoing treatment is not exclusionary (for example packed red blood cells emergently given during an elective surgery).
18. Receipt of another investigational agent within 3 months prior to viral inoculation.
19. Individual with body mass index (BMI) less than or equal to 18.5 or greater than or equal to 37.5.
20. Any significant abnormality of the nose or nasopharynx, including recurrent epistaxis within 3 months prior to viral inoculation.
21. Nasal or sinus surgery within 6 months prior to viral inoculation.
22. Shares household, works closely with, or has routine contact with a child (children) < 5 years of age or with immunocompromised individual(s), adults with significant cardiopulmonary disease, persons with significant asthma, institutionalized elderly or elderly with functional disability or any other individual that, in the judgment of the PI, might be at increased risk for complications if exposed to RSV.
23. Deprived of freedom by an administrative or court order or in an emergency setting.
24. Any condition that in the opinion of the principal investigator (PI) would jeopardize the safety or rights of a person participating in the trial or would render the person unable to comply with the protocol.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2015-07-21 (Actual); Primary Completion 2016-08-10 (Actual); Study Completion 2016-08-10 (Actual)

PRIMARY OUTCOMES:
Collection and assessment of expected and unexpected AEs. | Safety will be assessed continuously during inpatient and outpatient phases of the study through Day 56
  Safety

SECONDARY OUTCOMES:
RSV challenge associated viral shedding from nasal secretions: viral titer onset, duration, peak, and AUC | Viral shedding was assessed daily during the inpatient phase starting on day 2 following virus inoculation through day of discharge
  Viral shedding detected in nasal wash
RSV challenge associated immune responses: neutralizing antibody and immune cell phenotyping | Immune responses were assessed on days -1, 1, 7, and 10 during inpatient stay. Immune response were also examined during outpatient visits on day 28, day 56, and day 180.
  Antibody and T cell responses
RSV challenge associated clinical disease: frequency of upper respiratory infection, symptom score, and mucous weights | Clinical signs and symptoms were assessed daily during the inpatient phase. Interim history and physical was performed during outpatient visits.
  RSV Illness

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey I Cohen, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Lee FE, Walsh EE, Falsey AR, Betts RF, Treanor JJ. Experimental infection of humans with A2 respiratory syncytial virus. Antiviral Res. 2004 Sep;63(3):191-6. doi: 10.1016/j.antiviral.2004.04.005. PMID 15451187
- [Background] DeVincenzo JP, Wilkinson T, Vaishnaw A, Cehelsky J, Meyers R, Nochur S, Harrison L, Meeking P, Mann A, Moane E, Oxford J, Pareek R, Moore R, Walsh E, Studholme R, Dorsett P, Alvarez R, Lambkin-Williams R. Viral load drives disease in humans experimentally infected with respiratory syncytial virus. Am J Respir Crit Care Med. 2010 Nov 15;182(10):1305-14. doi: 10.1164/rccm.201002-0221OC. Epub 2010 Jul 9. PMID 20622030
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-I-0148.html